CLINICAL TRIAL: NCT04751058
Title: Genetic Profile in Patients With Aortic Syndrome
Acronym: GEN-AOR
Status: Completed | Type: Observational
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Antonio M. Puppo Moreno, Principal Investigator, Hospitales Universitarios Virgen del Rocío
Other Study IDs: HU Virgen Rocio
Record Dates: First submitted 2020-12-21; First posted 2021-02-11 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Gene Abnormality; Acute Aortic Syndrome
MeSH Terms: conditions — Acute Aortic Syndrome | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: genetic analysis — Intervention details: sampling in peripheral blood for the Methodology:
  1. Automatic DNA extraction (ChemagicTM 360)
  2. Mass sequencing using SeqCap EZ Choice Library capture technology (NimbleGen) and NextSeq sequencer (Illumina).
  3. Bioinformatic analysis:.
     * Identification of point mutations and small deletions or insertions
     * Analysis of CNVs using the BEDtools program package
     * Search of the identified variants in the following public databases: 1000G, dbSNP, ExAC, EVS, GenomADm CSVS and DGV. Those with a MAF> 1% have been considered benign, in public or private databases of our population.
  The analysis process has focused exclusively on the genes described to date as associated with the pathology under study and included in the panel used. The reference sequences used for these genes are: determination of possible mutations, nucleotics, etc.

SUMMARY:
The overall prevalence has increased significantly in the general population, which may be due in part to advances in diagnostic techniques, such as improved imaging techniques. Aortic dissection (AD) can cause sudden cardiac death (SCD). Approximately 95% of thoracic AAS are clinically "silent" until a life-threatening complication arises in an unpredictable manner and presents as sudden cardiac death. The peak incidence of death caused by aortic dissection occurs within 48 hours, therefore, timely diagnosis is essential and saves lives.

We have traditionally associated as risk factors in patients with ASA long-term arterial hypertension, present in 66-75% of cases, smoking, dyslipidemia or atherosclerotic disease. Likewise, any condition that alters the structure of the aorta such as: collagen diseases, aneurysms, bicuspid aorta, and manipulation of the thoracic aorta (cardiac surgery, 18%, or percutaneous intervention that can injure the intima) is involved in ASA. In addition to the well-known hereditary syndromes that affect collagen (Marfan, Elher-Danlos ...) there is a clear familial aggregation: 13-19% of patients without identifiable syndrome have first-degree relatives with thoracic aortic aneurysms or ICD, something that has been called "thoracic aortic dissection and familial aneurysm syndrome."

Notable achievements have been made in the discovery of genetic mutations associated with SAA and key regulatory molecules involved, including the extracellular matrix (ECM), cytoskeletal proteins, and the TGF-β signaling pathway. Identification of the causative gene is advantageous for both patients and their families, especially those who do not show symptoms. The specific underlying genotype could benefit the process of diagnosis, surveillance and surgery, with the aim of reducing morbidity and mortality

DETAILED DESCRIPTION:
HYPOTHESIS.:

A proportion of patients admitted to the Hospital with a diagnosis of Aortic Syndrome without phenotypic characteristics are carriers of mutations. The presence of these mutations can condition both the indication for treatment, post-surgical aortic remodeling, and family traceability.

OBJECTIVE.:

The objective of this study is to analyze the prevalence of mutations in non-phenotypic patients admitted urgently due to Aortic Syndrome.

Material and method:

Patients admitted to the Intensive Care Unit of the Virgen del Rocio University Hospital in Seville (third level Hospital) with the diagnosis of Aortic Syndrome will be included. The clinical and angiographic variables were analyzed. All patients will undergo, with prior informed consent, a peripheral blood extraction, from which a DNA sample will be obtained using the ChemagicTM 360 equipment. This DNA will be processed for massive sequencing on Illumina's NextSeq500 platform using the technology Capture SeqCap EZ Choice Library NimbleGen. The data generated will be analyzed bioinformatically and the identified variants prioritized based on their population frequency (<0.01), location (exonic and close to splicing sites), their presence in databases of clinical significance ClinVar, HGMD and LOVD and the phenotypic association of the mutated gene OMIM and Orphanet.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 16 years
* Patients admitted alive with a diagnosis of acute aortic syndrome
* Written consent to be DNA analysis and conservation in the DNA bank

Exclusion Criteria:

* Refusal to participate in the study and , or analysis of their DNA.
* Without life expectancy and , or Income without life.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study includes all patients who are admitted with the diagnosis of Acute Aortic Syndrome verified by imaging techniques (CT Angiography) in the Intensive Care Unit of a tertiary Hospital with a 24-hour Cardiac and Vascular Surgery Service
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-02-27 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
% of patients with presence of Missense mutations | post-treatment
  massive sequencing
% of patients with presence of splicing mutations | post-treatment
  massive sequencing
% of patients with presence of frameshift mutations | post-treatment
  massive sequencing
% of patients with presence of nonframeshift mutations | post-treatment
  massive sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Antonio M Puppo Moreno, MD;PhD, Principal Investigator — Andaluz Health Service
Locations (2):
- Spain (2):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bravo-Gil N, Gonzalez-Del Pozo M, Martin-Sanchez M, Mendez-Vidal C, Rodriguez-de la Rua E, Borrego S, Antinolo G. Unravelling the genetic basis of simplex Retinitis Pigmentosa cases. Sci Rep. 2017 Feb 3;7:41937. doi: 10.1038/srep41937. PMID 28157192
- [Background] Lopez-Domingo FJ, Florido JP, Rueda A, Dopazo J, Santoyo-Lopez J. ngsCAT: a tool to assess the efficiency of targeted enrichment sequencing. Bioinformatics. 2014 Jun 15;30(12):1767-8. doi: 10.1093/bioinformatics/btu108. Epub 2014 Feb 26. PMID 24578402
- [Background] Biddinger A, Rocklin M, Coselli J, Milewicz DM. Familial thoracic aortic dilatations and dissections: a case control study. J Vasc Surg. 1997 Mar;25(3):506-11. doi: 10.1016/s0741-5214(97)70261-1. PMID 9081132
- [Background] Albornoz G, Coady MA, Roberts M, Davies RR, Tranquilli M, Rizzo JA, Elefteriades JA. Familial thoracic aortic aneurysms and dissections--incidence, modes of inheritance, and phenotypic patterns. Ann Thorac Surg. 2006 Oct;82(4):1400-5. doi: 10.1016/j.athoracsur.2006.04.098. PMID 16996941
- [Background] Coady MA, Davies RR, Roberts M, Goldstein LJ, Rogalski MJ, Rizzo JA, Hammond GL, Kopf GS, Elefteriades JA. Familial patterns of thoracic aortic aneurysms. Arch Surg. 1999 Apr;134(4):361-7. doi: 10.1001/archsurg.134.4.361. PMID 10199307
- [Background] Milewicz D, Hostetler E, Wallace S, Mellor-Crummey L, Gong L, Pannu H, Guo DC, Regalado E. Precision medical and surgical management for thoracic aortic aneurysms and acute aortic dissections based on the causative mutant gene. J Cardiovasc Surg (Torino). 2016 Apr;57(2):172-7. Epub 2016 Feb 2. PMID 26837258
- [Background] Elefteriades JA, Farkas EA. Thoracic aortic aneurysm clinically pertinent controversies and uncertainties. J Am Coll Cardiol. 2010 Mar 2;55(9):841-57. doi: 10.1016/j.jacc.2009.08.084. PMID 20185035
- [Background] Milewicz DM, Chen H, Park ES, Petty EM, Zaghi H, Shashidhar G, Willing M, Patel V. Reduced penetrance and variable expressivity of familial thoracic aortic aneurysms/dissections. Am J Cardiol. 1998 Aug 15;82(4):474-9. doi: 10.1016/s0002-9149(98)00364-6. PMID 9723636
- [Background] Robertson EN, van der Linde D, Sherrah AG, Vallely MP, Wilson M, Bannon PG, Jeremy RW. Familial non-syndromal thoracic aortic aneurysms and dissections - Incidence and family screening outcomes. Int J Cardiol. 2016 Oct 1;220:43-51. doi: 10.1016/j.ijcard.2016.06.086. Epub 2016 Jun 23. PMID 27372041
- [Background] Renner S, Schuler H, Alawi M, Kolbe V, Rybczynski M, Woitschach R, Sheikhzadeh S, Stark VC, Olfe J, Roser E, Seggewies FS, Mahlmann A, Hempel M, Hartmann MJ, Hillebrand M, Wieczorek D, Volk AE, Kloth K, Koch-Hogrebe M, Abou Jamra R, Mitter D, Altmuller J, Wey-Fabrizius A, Petersen C, Rau I, Borck G, Kubisch C, Mir TS, von Kodolitsch Y, Kutsche K, Rosenberger G. Next-generation sequencing of 32 genes associated with hereditary aortopathies and related disorders of connective tissue in a cohort of 199 patients. Genet Med. 2019 Aug;21(8):1832-1841. doi: 10.1038/s41436-019-0435-z. Epub 2019 Jan 24. PMID 30675029
- [Background] Poninska JK, Bilinska ZT, Franaszczyk M, Michalak E, Rydzanicz M, Szpakowski E, Pollak A, Milanowska B, Truszkowska G, Chmielewski P, Sioma A, Janaszek-Sitkowska H, Klisiewicz A, Michalowska I, Makowiecka-Ciesla M, Kolsut P, Stawinski P, Foss-Nieradko B, Szperl M, Grzybowski J, Hoffman P, Januszewicz A, Kusmierczyk M, Ploski R. Next-generation sequencing for diagnosis of thoracic aortic aneurysms and dissections: diagnostic yield, novel mutations and genotype phenotype correlations. J Transl Med. 2016 May 4;14(1):115. doi: 10.1186/s12967-016-0870-4. PMID 27146836
- [Background] Proost D, Vandeweyer G, Meester JA, Salemink S, Kempers M, Ingram C, Peeters N, Saenen J, Vrints C, Lacro RV, Roden D, Wuyts W, Dietz HC, Mortier G, Loeys BL, Van Laer L. Performant Mutation Identification Using Targeted Next-Generation Sequencing of 14 Thoracic Aortic Aneurysm Genes. Hum Mutat. 2015 Aug;36(8):808-14. doi: 10.1002/humu.22802. Epub 2015 Jun 13. PMID 25907466
- [Background] Arslan-Kirchner M, Arbustini E, Boileau C, Charron P, Child AH, Collod-Beroud G, De Backer J, De Paepe A, Dierking A, Faivre L, Hoffjan S, Jondeau G, Keyser B, Loeys B, Mayer K, Robinson PN, Schmidtke J. Clinical utility gene card for: Hereditary thoracic aortic aneurysm and dissection including next-generation sequencing-based approaches. Eur J Hum Genet. 2016 Jan;24(1):e1-5. doi: 10.1038/ejhg.2015.225. Epub 2015 Oct 28. No abstract available. PMID 26508578
- [Background] Renard M, Francis C, Ghosh R, Scott AF, Witmer PD, Ades LC, Andelfinger GU, Arnaud P, Boileau C, Callewaert BL, Guo D, Hanna N, Lindsay ME, Morisaki H, Morisaki T, Pachter N, Robert L, Van Laer L, Dietz HC, Loeys BL, Milewicz DM, De Backer J. Clinical Validity of Genes for Heritable Thoracic Aortic Aneurysm and Dissection. J Am Coll Cardiol. 2018 Aug 7;72(6):605-615. doi: 10.1016/j.jacc.2018.04.089. PMID 30071989
- [Background] Zheng J, Guo J, Huang L, Wu Q, Yin K, Wang L, Zhang T, Quan L, Zhao Q, Cheng J. Genetic diagnosis of acute aortic dissection in South China Han population using next-generation sequencing. Int J Legal Med. 2018 Sep;132(5):1273-1280. doi: 10.1007/s00414-018-1890-9. Epub 2018 Jul 28. PMID 30056620
- [Background] Arnaud P, Hanna N, Benarroch L, Aubart M, Bal L, Bouvagnet P, Busa T, Dulac Y, Dupuis-Girod S, Edouard T, Faivre L, Gouya L, Lacombe D, Langeois M, Leheup B, Milleron O, Naudion S, Odent S, Tchitchinadze M, Ropers J, Jondeau G, Boileau C. Genetic diversity and pathogenic variants as possible predictors of severity in a French sample of nonsyndromic heritable thoracic aortic aneurysms and dissections (nshTAAD). Genet Med. 2019 Sep;21(9):2015-2024. doi: 10.1038/s41436-019-0444-y. Epub 2019 Feb 11. PMID 30739908
- [Background] Clouse WD, Hallett JW Jr, Schaff HV, Spittell PC, Rowland CM, Ilstrup DM, Melton LJ 3rd. Acute aortic dissection: population-based incidence compared with degenerative aortic aneurysm rupture. Mayo Clin Proc. 2004 Feb;79(2):176-80. doi: 10.4065/79.2.176. PMID 14959911
- [Background] Meszaros I, Morocz J, Szlavi J, Schmidt J, Tornoci L, Nagy L, Szep L. Epidemiology and clinicopathology of aortic dissection. Chest. 2000 May;117(5):1271-8. doi: 10.1378/chest.117.5.1271. PMID 10807810
- [Background] Kuzmik GA, Sang AX, Elefteriades JA. Natural history of thoracic aortic aneurysms. J Vasc Surg. 2012 Aug;56(2):565-71. doi: 10.1016/j.jvs.2012.04.053. PMID 22840907
- [Background] Gago-Diaz M, Ramos-Luis E, Zoppis S, Zorio E, Molina P, Braza-Boils A, Giner J, Sobrino B, Amigo J, Blanco-Verea A, Carracedo A, Brion M. Postmortem genetic testing should be recommended in sudden cardiac death cases due to thoracic aortic dissection. Int J Legal Med. 2017 Sep;131(5):1211-1219. doi: 10.1007/s00414-017-1583-9. Epub 2017 Apr 8. PMID 28391405
- [Background] Erbel R, Aboyans V, Boileau C, Bossone E, Bartolomeo RD, Eggebrecht H, Evangelista A, Falk V, Frank H, Gaemperli O, Grabenwoger M, Haverich A, Iung B, Manolis AJ, Meijboom F, Nienaber CA, Roffi M, Rousseau H, Sechtem U, Sirnes PA, Allmen RS, Vrints CJ; ESC Committee for Practice Guidelines. 2014 ESC Guidelines on the diagnosis and treatment of aortic diseases: Document covering acute and chronic aortic diseases of the thoracic and abdominal aorta of the adult. The Task Force for the Diagnosis and Treatment of Aortic Diseases of the European Society of Cardiology (ESC). Eur Heart J. 2014 Nov 1;35(41):2873-926. doi: 10.1093/eurheartj/ehu281. Epub 2014 Aug 29. No abstract available. PMID 25173340
- [Derived] Puppo Moreno AM, Bravo-Gil N, Mendez-Vidal C, Adsuar Gomez A, Gomez Ruiz FT, Jimenez De Juan C, Fernandez Garcia RM, Martin Bermudez R, Lopez Sanchez JM, Martin Sastre S, Fernandez Caro M, Gallego P, Borrego S. Genetic profile in patients with complicated acute aortic syndrome: the GEN-AOR study. Rev Esp Cardiol (Engl Ed). 2023 Jun;76(6):434-443. doi: 10.1016/j.rec.2022.10.005. Epub 2022 Oct 25. English, Spanish. PMID 36307044